CLINICAL TRIAL: NCT01960634
Title: Translational Study for BRAFV600 Serum and Plasma Determination in Patients With BRAFV600 Metastatic Melanoma
Acronym: BRAFV600
Status: Completed | Type: Observational
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Responsible Party: Sponsor
Other Study IDs: GEM-1304; GEM-1304 (Other: Sponsor)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-centric translational study with biological samples collection. The aim of this study is to validate a method to detect BRAFV600 in blood samples.

Samples: Blood from patients with BRAFV600 metastatic melanoma collected following standard medical practice.

The treatment is not the aim of the study. Patients can be treated either with specific or no-specific drug.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of melanoma and BRAFV600
* Signed Informed Consent Form
* Unresectable phase III or phase IV melanoma
* The patients should be starting a treatment for melanoma (either first line or subsequent lines)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed melanoma and BRAF V600 mutation
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Rate of patient in which BRAF V600 in blood samples is present/absent | two years

SECONDARY OUTCOMES:
Rate of patients with BRAFV600 present in tumor sample vs blood sample | two years

OTHER OUTCOMES:
BRAF V600 blood levels and illness evolution | two years
NRAS and p61BRAFFV600 serum levels and clinic evolution | two years
BRAFV600 blood levels vs progression-free survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: María González Cao, MD, Study Director — Hospital Universitario Quirón Dexeus
Locations (13):
- Spain (13):
  - Hospital Infanta Cristina, Madrid, Badajoz
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario Quirón Dexeus, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Costa del SOl, Marbella, Málaga
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza, Zaragoza